CLINICAL TRIAL: NCT03090438
Title: The Effect of Preliminary Varicocele Repair on IVF Outcomes in Male Factor Infertility
Brief Title: IVF Outcomes After Varicocele Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZMCvarivf
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2016-10

CONDITIONS: Infertility, Male; Varicocele; In Vitro Fertilization
MeSH Terms: conditions — Infertility, Male; Varicocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Varicocele embolization before IVF (Active Comparator): Participants will have catheterization and embolization of varicoceles six months before beginning IVF
  Interventions: Procedure: Varicocele embolization
- IVF without varicocele embolization (No Intervention): Participants will proceed from enrollment directly to IVF

INTERVENTIONS:
Procedure: Varicocele embolization — Ultrasound guided right internal jugular vein access with placement of a vascular sheath. Fluoroscopically guided selective catheterization of the left and right (if bilateral) spermatic veins to the level of the inguinal ligament. Occlusion of the spermatic vein(s) by embolization coils and a sclerosing agent (sodium tetradecyl sulphate 3%).
  Other Names: Varicocele repair; Varicocele occlusion
  Arms: Varicocele embolization before IVF

SUMMARY:
Infertility has been estimated to affect from 6-18% of couples trying to conceive. In 20-30% of cases, the problem is with the male. Varicocele is a common cause of male factor infertility (MFI) being responsible for 30-35 % of primary and 69-81 % of secondary MFI. Varicocele repair has been shown to improve sperm parameters and increase natural pregnancy rates and the results of assisted reproductive techniques (ART).

There are two possible treatment pathways for varicocele associated male factor infertility. 1) standard IVF/ICSI 2) varicocele repair followed by IVF/ICSI if there is no spontaneous pregnancy. There is however no consensus as to which pathway is preferable and no randomized comparative studies have been carried out.

IVF/ICSI is a standard treatment for infertility but frequently requires repeated treatments to achieve a live birth. The purpose of this study is to determine if the improved sperm parameters caused by prior treatment of the varicocele will result in improvements both in overall pregnancy/birth rates and in IVF/ICSI results.

DETAILED DESCRIPTION:
A varicocele is an abnormal dilation of the pampiniform plexus caused by incompetence of the valves in the internal spermatic vein. Varicocele has a prevalence of 10-15 % in the general population and is a common cause of male infertility, being present in 30-35% of men with primary, and 69-81% of men with secondary infertility. There is more than one approach to the treatment of varicocele associated MFI One common approach is to treat by assisted reproductive techniques (ART). Patients with a total motile sperm count of <10 million sperm are usually treated by IVF with or without ICSI. Fertilization of oocytes may be accomplished by isolating even a single adequate spermatozoa in the laboratory bypassing the majority of semen quality inadequacies in male factor infertility. The results of this treatment using fresh embryos with a maternal age of<35 are 46% pregnancies and 40% live births per cycle.

Alternatively, varicocele associated MFI can be treated by repairing the varicocele to improve sperm quality. Occlusion of the spermatic veins by surgical and radiological methods is commonly performed in these circumstances to improve fertility. A large body of literature exists demonstrating post-treatment improvements in semen parameters and sperm DNA quality as well as improved spontaneous pregnancy rates compared to no treatment. There are also studies demonstrating improved results of ART after varicocele repair.

Both approaches have their advocates. ART often provide a relatively quick result and have a known excellent track record for both pregnancy and live birth rates. Unfortunately, these techniques are not without risks such as ovarian hyperstimulation syndrome and procedural complications. Multiple pregnancies are common with increased risk of premature labour and low birth weight. In addition the treatments are expensive and multiple treatments increase the financial burden on the health care system.

Varicocele occlusion is a minor procedure. If performed radiologically, there is often immediate return to normal activity. The complication rate is very low, mostly due to radiological contrast medium allergy. Modern equipment and careful technique enable the procedure to be completed with very low radiation doses that are well below the level proven to have any adverse biological effect.

If varicocele repair can be demonstrated to improve pregnancy outcomes in varicocele related MFI by spontaneous pregnancies or by improving pregnancy and live birth rates per ART implantation, then there are compelling health care and economic reasons for incorporating it as an initial treatment.

At present there have been no well constructed randomized trials to compare the outcomes of these two approaches.

ELIGIBILITY:
Inclusion Criteria:

Patient complies to varicocele treatment indications as per ASRM 2014 guidelines

1. Palpable varicocele on physical exam
2. The female partner has normal fertility or a potentially treatable cause of infertility
3. Male has abnormal semen parameters

Age of female partner < 35 years

Exclusion Criteria:

Sub-clinical varicocele

Isolated teratospermia

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 25 months
  The percentage of embryo transfers resulting in a live birth

SECONDARY OUTCOMES:
Pregnancy rate | 18 months
  The percentage of embryo transfers resulting in a clinical pregnancy ((ultrasound visualization of a gestational sac with heartbeat)
Transfers per clinical pregnancy | 18 months
  Total transfers divided by total clinical pregnancies (excluding natural pregnancies) for each study group
Transfers per live birth | 25 months
  Total transfers divided by total live births (excluding natural pregnancies) for each study group
Ongoing pregnancy rate | 18 months
  Number of pregnancies (including natural) at 3 month time intervals
Ongoing live birth rate | 25 months
  Number of live births (including natural) at 3 month time intervals

CONTACTS AND LOCATIONS:
Overall Officials: Anthony G Verstandig, MD, Principal Investigator — C; Ruth Ronn, MD, Principal Investigator — V

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorelick JI, Goldstein M. Loss of fertility in men with varicocele. Fertil Steril. 1993 Mar;59(3):613-6. PMID 8458466
- [Background] Agarwal A, Deepinder F, Cocuzza M, Agarwal R, Short RA, Sabanegh E, Marmar JL. Efficacy of varicocelectomy in improving semen parameters: new meta-analytical approach. Urology. 2007 Sep;70(3):532-8. doi: 10.1016/j.urology.2007.04.011. PMID 17905111
- [Background] Diegidio P, Jhaveri JK, Ghannam S, Pinkhasov R, Shabsigh R, Fisch H. Review of current varicocelectomy techniques and their outcomes. BJU Int. 2011 Oct;108(7):1157-72. doi: 10.1111/j.1464-410X.2010.09959.x. Epub 2011 Mar 24. PMID 21435155
- [Background] Verstandig AG, Shamieh B, Shraibman V, Raveh D. Radiation dose reduction in fluoroscopic procedures: left varicocele embolization as a model. Eur Radiol. 2015 Jun;25(6):1639-45. doi: 10.1007/s00330-014-3556-4. Epub 2014 Dec 19. PMID 25523457
- [Background] Esteves SC, Roque M, Agarwal A. Outcome of assisted reproductive technology in men with treated and untreated varicocele: systematic review and meta-analysis. Asian J Androl. 2016 Mar-Apr;18(2):254-8. doi: 10.4103/1008-682X.163269. PMID 26510504
- [Background] Kim KH, Lee JY, Kang DH, Lee H, Seo JT, Cho KS. Impact of surgical varicocele repair on pregnancy rate in subfertile men with clinical varicocele and impaired semen quality: a meta-analysis of randomized clinical trials. Korean J Urol. 2013 Oct;54(10):703-9. doi: 10.4111/kju.2013.54.10.703. Epub 2013 Oct 15. PMID 24175046
- [Background] Schauer I, Madersbacher S, Jost R, Hubner WA, Imhof M. The impact of varicocelectomy on sperm parameters: a meta-analysis. J Urol. 2012 May;187(5):1540-7. doi: 10.1016/j.juro.2011.12.084. Epub 2012 Mar 14. PMID 22425089
- [Background] Li F, Yamaguchi K, Okada K, Matsushita K, Ando M, Chiba K, Yue H, Fujisawa M. Significant improvement of sperm DNA quality after microsurgical repair of varicocele. Syst Biol Reprod Med. 2012 Oct;58(5):274-7. doi: 10.3109/19396368.2012.692431. Epub 2012 Jul 2. PMID 22979920
- [Background] The influence of varicocele on parameters of fertility in a large group of men presenting to infertility clinics. World Health Organization. Fertil Steril. 1992 Jun;57(6):1289-93. PMID 1601152